CLINICAL TRIAL: NCT04342338
Title: Pharmacist and Family Medicine Physician Collaboration for Pre-Visit Planning and Team Huddles for Patients Receiving Chronic Care Management Services
Brief Title: Pharmacist and Family Medicine Physician Collaboration for Pre-Visit Planning and Team Huddles for CCM Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Northeast Iowa Medical Education Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-003
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Chronic Conditions, Multiple
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a novel project which incorporates clinic and community pharmacists in three aspects of the Patient-Centered Medical Home: pre-visit planning, pre-visit care team huddles, and chronic care management (CCM). Patients for the project are enrolled in the NEIFPC CCM program and have Greenwood pharmacy as their primary pharmacy. Community and clinic pharmacists will contribute to pre-visit medication reviews and document their drug therapy recommendations in a shared, templated note in the clinic EHR. NEIFPC pharmacists will attend pre-visit team huddles to relay drug therapy recommendations to the physician. Revenue from CCM services will be prorated and shared between Greenwood pharmacy and NEIFPC. The project will last 9 months. Primary aims are to describe the pharmacist pre-visit planning service, summarize the billing experience of a community pharmacist providing this service, and to describe the drug therapy interventions made by pharmacists.

ELIGIBILITY:
Inclusion Criteria:

* Patient enrolled in Medicare
* Patient enrolled in the Chronic Care Management (CCM) program at the Northeast Iowa Family Practice Center
* Patient's primary pharmacy is Greenwood Pharmacy

Exclusion Criteria:

* Patient not enrolled in Medicare
* Patient not enrolled in CCM program
* Patient's primary pharmacy is any pharmacy other than Greenwood Pharmacy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Medicare patient's who are enrolled in the CCM program at the Northeast Iowa Family Practice Center with Greenwood Pharmacy as their primary pharmacy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Summary of Drug Therapy Interventions made by Pharmacists | 07/01/2020- 03/31/2021
  Summarize drug therapy interventions made by community and ambulatory care pharmacists for pre-visit team huddles with Family Medicine physicians.

CONTACTS AND LOCATIONS:
Locations (1):
- Northeast Iowa Family Practice, Waterloo, Iowa, United States